CLINICAL TRIAL: NCT00455364
Title: Assessment of Safety and Efficacy of Voriconazole as Prophylactic Antifungal Therapy for Lung Transplant Recipients
Brief Title: Voriconazole as Prophylactic Therapy in Lung Transplant Recipients
Acronym: VORI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Protocol never received funding.
Sponsor: University of Chicago (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14559A
Record Dates: First submitted 2007-04-02; First posted 2007-04-03 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Infection
Keywords: Fungal infection prophylaxis; Lung transplant; Fungal infection post lung transplant
MeSH Terms: conditions — Infections | interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Voriconazole

SUMMARY:
The purpose of this study is to compare the safety and efficacy of Voriconazole with Itraconazole following lung transplantation.

DETAILED DESCRIPTION:
All participants will receive itraconazole during their inpatient post transplant stay. As an outpatient, ten subjects will be randomized to receive itraconazole 200mg orally once daily for 6 month and ten patients to receive voriconazole 200mg orally twice daily for 6 months . All subjects will be followed in the clinic as per the standard transplant treatment

ELIGIBILITY:
Inclusion Criteria:

* Bilateral-lung or single-lung transplant recipients between the ages of 18- 65 years old.
* Patients must be able to give informed consent prior to and again after transplantation

Exclusion Criteria:

* Lung transplant patients unable to give informed consent.
* Prior adverse reaction to the drug itraconazole or voriconazole

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Subject will be monitored for any fungal infection throughout the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta Bhorade, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States